CLINICAL TRIAL: NCT01600781
Title: Effect of Oral Supplementation With a Fibre Enriched Paediatric Sip Feed on the Nutritional Status, Gut Microbiota and Quality of Life of Children With Acute Lymphocytic Leukemia: an Egyptian Pilot Study
Brief Title: Effect of Oral Supplementation With a Fibre Enriched Paediatric Sip Feed For Children With Acute Lymphocytic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCHE-ALL001
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: Improve the nutritional status; QOL; children; enhance immune response; induction chemotherapy; fewer side effects
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NutriniDrink/Fortini group (Active Comparator): this group will receive 2 bottles of NutriniDrink/Fortini MF unflavoured daily (200 ml each) and standard dietary counselling for a period of 6 weeks.
  Interventions: Dietary Supplement: NutriniDrink/Fortini MF unflavoured (1.5kcal/ml)
- control group (No Intervention): this control group will only receive standard dietary counselling

INTERVENTIONS:
Dietary Supplement: NutriniDrink/Fortini MF unflavoured (1.5kcal/ml) — During the 6-week Intervention period children allocated to group 1 will consume 2 bottles of study product per day (400ml in total).
  Arms: NutriniDrink/Fortini group

SUMMARY:
This is a randomised, controlled, open-label intervention study. It is hypothesized that supplementation with a fibre enriched sip feed will improve the nutritional status, gut microbiota and quality of life (QOL) of children with acute lymphoblastic leukemia, and may enhance their immune response. This could give them a better chance to finish their induction chemotherapy successfully with fewer side effects.

DETAILED DESCRIPTION:
Study objectives:

Primary objective:

To evaluate the effect of oral supplementation with a fibre supplemented paediatric sip feed on the nutritional status of Egyptian children with acute lymphocytic leukemia (ALL) compared to standard dietary counseling.

Secondary objective:

To evaluate the effect of oral supplementation with a fibre supplemented paediatric sip feed on the gut microbiota and quality of life (QoL) of Egyptian children with ALL compared to standard dietary counseling.

ELIGIBILITY:
Inclusion Criteria:• Newly diagnosed male and female paediatric ALL patients presenting in the study period.

* Age should be above 2 years and children should be pre-pubertal.
* Hospitalized for the entire (6 week) intervention period.
* About to receive? induction chemotherapy.
* Able to tolerate oral feeding.
* Written informed consent from parents/guardian (and child, if applicable to local law).

Exclusion Criteria:

* ALL patients < 2 years and those who show signs of puberty.
* ALL patients who cannot tolerate oral feeding and/or are on parenteral nutrition.
* ALL patients with a known history of cow's milk allergy/intolerance or galactosemia.
* ALL patients requiring a fibre-free diet.
* Investigator's uncertainty about the willingness or ability of the child/carer to comply with the protocol requirements.
* Participation in any other study involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Study Parameters | 42 days
  Primary
  * Change in body weight between Baseline and Day 42 [kg, weight-for-age z score, weight-for-height z-score]
  * Percentage of children with body weight loss between Baseline and Day 42 [%]

SECONDARY OUTCOMES:
Study Parameters | from day 1 to day 91 of the study
  * Stool microbiota at Baseline and at Day 42 [proportion of Bifidobacteria, total stool culture]
  * Quality of life at Baseline, at Day 42 and Day 91 [PedsQL Cancer Module]
  * Change in body weight between Baseline and Day 91 [kg, weight-for-age z score, weight-for-height z-score]
  * Percentage of children with body weight loss between Baseline and Day 91 [%]

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El-Hadad, PhD, Principal Investigator — Children's Cancer Hospita Egypt-57357
Locations (1):
- Children's cancer Hospital Egypt-57357, Cairo, Egypt